CLINICAL TRIAL: NCT05006963
Title: Tele-Rehabilitation in Patients With Temporomandibular Dysfunction: Randomized, Controlled and Blind
Brief Title: Tele-Rehabilitation in Patients With Temporomandibular Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, PhD, professor and researcher, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tele-Reabilitação em TMD
Record Dates: First submitted 2020-11-26; First posted 2021-08-16 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Disorder; Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome
Keywords: temporomandibular joint disorders; clinical protocols; physiotherapy; remote consultation; telemedicine; telehealth; telerehabilitation; teletherapy; telepractice
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Two researchers will be part of the protocol. One will be responsible for pre and post intervention assessments and will be blind to the type of intervention. The other will be responsible for the treatment phase: face-to-face and telerehabilitation. A third party collaborator will process and statistically analyze the collected data. Individuals will be randomized using the statistical program present at www.randomization.com , in two groups. Randomization and concealment of allocation will be made by a fourth external employee, not research participant, who will organize the allocation in individual opaque envelopesand keep it confidential. There will be 2 blocks of 25 envelopes: face-to-face (GA) and telerehabilitation (GB). With this process, participants will have the same probability of being allocated to one of the two treatment groups. Blinding of the evaluator will be maintained until the end of the research and data tabulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face-to-face group (Experimental): The patient will be submitted to multimodal treatment, twice a week, for twelve weeks, totaling 24 face-to-face consultations lasting 40 minutes each. In the first session, the patient will be explained what is TMD, what is the correct placement of the tongue and teeth, influence of parafunctional and sleep habits in TMD signs and symptoms.Techniques of manual therapy and therapy by exercise. In general, extra-oral and intraoral massage, myofascial release in the cranio-cervical musculature, mobilization of the hyoid bone and may also receive unspecific joint mobilization. Will be mouth opening exercise will be also performed with the tongue on the palate, proprioceptive exercises with hyperboloid. In addition to these, additional exercises may be performed, according to the patient's need. The conducts will be adapted according to the needs of each patient. The use of post its may be indicated to help maintain the correct posture of the tongue and jaw, as well as sleep hygiene.
  Interventions: Other: manual therapy and therapy by exercise
- telerehabilitation (Active Comparator): The patient will be submitted to multimodal treatment, twice a week, for twelve weeks, by telerehabilitation lasting 40 minutes each.A physiotherapist through video call via WhatsApp application. In the first session, the patient will be explained what is TMD, what is the correct placement of the tongue and teeth, influence of parafunctional and sleep habits in TMD signs and symptoms. Patients will be instructed to perform extra-oral and intra-oral self-massage and in the cranio-cervical musculature, bone mobilization hyoid, which would replace the mobilization unspecific articulation performed in person.Exercise will also be carried out mouth opening with tongue on the palate, exercises proprioceptives with hyperboloid. The conducts will be adapted according to the needs of each patient.The conducts will be adapted according to the needs of each patient.The use of post its may be indicated to help maintain the correct posture of the tongue and jaw, as well as sleep hygiene
  Interventions: Other: manual therapy and therapy by exercise

INTERVENTIONS:
Other: manual therapy and therapy by exercise — In general, patients will receive extra-oral massage and intraoral massage, myofascial release in the cranio-cervical musculature, mobilization of the hyoid bone and may also receive unspecific joint mobilization. Will bemouth opening exercise was also performed with the tongue on the palate, proprioceptive lateralization and protrusion exercises with hyperboloid and exercises with combinations of movements of laterality and opening, or protrusion and opening.

SUMMARY:
Temporomandibular disorder or TMD is characterized by a set of symptoms such as: pain, decreased range of motion and joint noise. It's origin is multifactorial, which may be related to biological aspects, environmental and psychosocial. The multimodal approach has been widely used in physiotherapy for the treatment of TMDs. Physiotherapy has been walking together with technology so that telerehabilitation can be a reality, contributing so that quality care reaches the patient, in the impossibility office-to-face service. The objective of this study is to verify the effect of telerehabilitation on pain outcomes, range of motion, functionality and biopsychosocial aspects in individuals with temporomandibular disorders. Will be a randomized, controlled and blinded clinical trial was carried out. The study will be divided into two moments: evaluation and intervention. Evaluations will be carried out using the Diagnostic Criteria for Temporomandibular Disorders: Clinical Protocol and Assessment Instruments (DC/TMD), the Fonseca Anamnesis Index (IAF), the Numerical Pain Scale (END) and the Functional Limitation Questionnaire (MFIQ). Individuals will be randomized into 2 groups: Group A (in person) Group B (telerehabilitation). Both groups will receive treatment physical therapy for 12 weeks. After collecting the data, they will be tabulated and analyzed using a 5% significance level.

ELIGIBILITY:
1. Age between 18 and 60 years;
2. presence of pain in the facial region in the last 6 months;
3. diagnosis of myalgia, arthralgia, headache attributed to temporomandibular disfunction and/or subluxation temporomandibular joint.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Score in Numerical Pain Scale | The level of pain at 12 weeks
  intensity of pain
Score in Numerical Pain Scale | The level of pain at 6 months
  intensity of pain
measure range of motion | The range of motion at range of motion at 12 weeks .
  range of motion
measure range of motion | The range of motion at 6 months.
  range of motion

SECONDARY OUTCOMES:
measure Functionality | The functionality at 12 weeks .
  Mandibular Functional Limitation Questionnaire
measure Functionality | The functionality at 6 months.
  Mandibular Functional Limitation Questionnaire
Biopsychosocial analysis. | The biopsychosocial analysis at 12 weeks .
  Axis II of the diagnostic criterion for temporomandibular disorders
Biopsychosocial analysis. | The biopsychosocial analysis at 6 months.
  Axis II of the diagnostic criterion for temporomandibular disorders

CONTACTS AND LOCATIONS:
Locations (1):
- University Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data is confidential, but if any journal requests open data for publication for sure we will provide our database